CLINICAL TRIAL: NCT06495554
Title: The Value of Patient-reported Outcome Measure Assessment and Circulating Tumor-DNA to Detect Early Relapse During Surveillance in Women With Vulva Cancer
Brief Title: Danish Vulva Cancer Recurrence Study
Acronym: DaVulvaRec
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Danish Cancer Society (Other); Danish Comprehensive Cancer Center (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1-10-72-150-23
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Vulva Cancer; Vulva Neoplasm; Vulvar Cancer; Vulva Disease; Vulvar Neoplasms; Vulvar Diseases; PROM; Circulating Tumor DNA; Survivorship
MeSH Terms: conditions — Vulvar Neoplasms; Vulvar Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROM assessment and ctDNA detection during surveillance (Experimental): All participants (n=295) included in the prospective clinical study
  Interventions: Diagnostic Test: Measurement of circulating tumor-DNA; Other: Collection of patient-reported outcomes; Other: Algorithmically determined telephone interview with a nurse
- Standard surveillance (No Intervention): Historical controls (n=1,000) who will be identified by the Danish Gynecological Cancer Database

INTERVENTIONS:
Diagnostic Test: Measurement of circulating tumor-DNA — Liquid biopsies will be collected at baseline and prospectively during follow-up to measure circulating tumor-DNA.
  Arms: PROM assessment and ctDNA detection during surveillance
Other: Collection of patient-reported outcomes — Patient-reported outcomes will be collected at baseline and prospectively during follow-up.
  Arms: PROM assessment and ctDNA detection during surveillance
Other: Algorithmically determined telephone interview with a nurse — Dependent on the patient's responses on the patient-reported outcome measures.
  Arms: PROM assessment and ctDNA detection during surveillance

SUMMARY:
The overall aim is to investigate different aspects of recurrence detection in women with vulva cancer (VC) to identify optimal treatment- and surveillance programs.

DaVulvaRec is a Danish nationwide multicenter study with patient inclusion from Aarhus University Hospital and Rigshospitalet, Denmark. Applying a mixed method research design, the investigators will collect and analyze patient-reported outcome measures in combination with procedural data to evaluate symptomatology and map actions taken during the patient's pathway from primary disease to recurrence. Furthermore, the investigators aim to examine if circulating tumor-DNA (ctDNA) can be detected in liquid biopsies from VC patients. All patients will be followed for two years or until recurrence. Patient-reported outcome measures will be completed every four months during surveillance, and liquid biopsies will be collected prospectively for later analyses.

Total number of patients to be included is 295 according to a power calculation. All patients in the clinical study will be included in the intervention group, while data on a historical control group will be obtained from The Danish Gynecological Cancer Database. Hence, the control group will consist of 1000 VC patients diagnosed between 2011-2022.

Hypotheses:

* All patients with VC will have specific tumor markers in the primary tumor that will be detectable in liquid biopsies as ctDNA at the time of diagnosis.
* Measurement of ctDNA after primary treatment and during surveillance will allow detection of residual disease, improve allocation for adjuvant treatment, and will allow early detection of recurrent VC.
* Proactive use of repeated PROM assessments in combination with procedural actions during surveillance will allow early detection of recurrent VC and early identification of late effects after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Primary or recurrent biopsy-verified squamous cell carcinoma of the vulva
* ≥ 18 years of age
* Able to understand oral and written information in Danish

Exclusion Criteria:

* Active treatment for concurrent cancer and/or dissemination of concurrent cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1295 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | Two years
Overall survival | Two years

SECONDARY OUTCOMES:
Symptomatology preceding a recurrence | Two years
Improved quality-of-life as a result of proactive management of late effects on an individual level | Two years
Improved survival as a result of proactive management of late effects on group level | Two years
ctDNA detection at time of diagnosis in relation to disease stage | Two years
ctDNA detection after end of treatment in relation to residual disease | Two years
ctDNA detection during surveillance in relation to recurrent disease | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Pernille T. Jensen, Professor, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Copenhagen University Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: No